CLINICAL TRIAL: NCT03295708
Title: Safety, Effectiveness, and Mechanism of Fish Oil as Adjunct Treatment for Major Depressive Disorder - a 12-month Randomized, Placebo Controlled Clinical Trial
Brief Title: Fish Oil as Adjunct Treatment for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jin-Dong Chen, Director of Mental Health Institute of the Second Xiangya Hospital, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDD201610
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder,Fish Oil
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): the experimental group will be given 4 fish oil capsules (1g/one capsule)twice daily after two meals at roughly the same time each day,lasting for the first 6 months.fish oil capsule will be provided by the Hunan Kangqi100 Biological Technology Co.Ltd.
  Interventions: Dietary Supplement: fish oil capsule
- control group (Placebo Comparator): the control group will be given 4 soybean oil capsules ( placebo capsule,1g/one capsule) twice daily after two meals at roughly the same time each day,lasting for the first 6 months.placebo capsule will be provided by the Hunan Kangqi100 Biological Technology Co.Ltd.The placebo capsule's appearance and flavor are made the exactly the same as the fish oil capsules .
  Interventions: Dietary Supplement: soybean oil capsule

INTERVENTIONS:
Dietary Supplement: fish oil capsule — N-3 PUFAs is a kind of essential fatty acid,however the formation is too slow. Studies show that intakes of N-3 PUFAs is associated with MDD.It have to be got from food like deep-sea fishes. EPA and DHA are crucial for the body.Although studies have shown that reduced N-3 PUFAs were correlated with MDD, and patients with an elevated rate of N-6 PUFAs /N-3 PUFAs or a low level of DHA may be at higher odds for suicide. Trials on whether N-3 PUFAs is effective in the treatment of MDD is still controversial, which might be affected by several factors, such as dose, duration etc.. Now there is no large-scale randomized controlled clinical trial in determining the effects of N-3 PUFAs add-on in treatment of MDD.
  Arms: experimental group
Dietary Supplement: soybean oil capsule — placebo capsule
  Arms: control group

SUMMARY:
In this proposed study, the investigators will evaluate the effects of fish oil add-on in treatment of major depressive disorder(MDD).

DETAILED DESCRIPTION:
Participants are randomly assigned to two groups (n=60): control (placebo, soybean) and fish oil (containing EPA 1440mg, DHA 960mg). The experimental groups will be compared to placebo to evaluate if it may benefit clinical symptoms, cognitive symptoms and metabolic markers in MDD patients. We also plan to investigate the changes in markers of inflammation at the same time.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Men or women aged 18-50 years
3. A primary psychiatric diagnosis of major depressive disorder (MDD), by Diagnostic and Statistical Manual-5th ed (DSM-5) using the MINI
4. HAMD total score≥21
5. No significantly modification of their diet from the time they sign consent to the end of study participation

Exclusion Criteria:

1. Suffering from other serious somatic diseases or comorbidities
2. Patients with serious nervous system disease
3. Patients in accordance with diagnostic standards of other mental illness
4. Patients who need to take benzodiazepine every day, and who currently need to be treated by electroconvulsive therapy or have received electroconvulsive therapy in the past 6 months
5. Pregnant women or lactating women, women with pregnancy plans during the trial period (12 months), women with a high risk of pregnancy but without taking any contraceptive measures
6. Patients with apparent suicide attempt or suicidal behavior
7. Any condition or medicines that may have an effect on biomarkers (within 1 week of the screening period or during whole trial period): long-term, regular use of NSAIDs, COX-2 inhibitors, immunosuppressant, steroids, interferon, chemotherapeutics, anticoagulants, malignancy, active autoimmune diseases, inflammatory bowel diseases, etc
8. Allergy history of PUFA
9. Intake of Fish oil more than 3g per day or eat fatty fish more than 3 times a week

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Hamilton Depression Scale (HAMD) HAMD | W0 W4 W12 W24 W48
  Subjects were evaluated for current depression with HAMD.

SECONDARY OUTCOMES:
Changes in Clinical Global Impression (CGI) | W0 W4 W12 W24 W48
  Subjects were evaluated for current severity of disease with CGI.
Changes in Hamilton Anxiety Scale (HAMA) | W0 W4 W12 W24 W48
  Subjects were evaluated for current anxiety with HAMA.
Changes in Beck Depression Rating Scale (BDI) | W0 W4 W12 W24 W48
  The BDI is a self-report inventory of depression symptom.
Changes in Self-Rating Anxiety Scale (SAS) | W0 W4 W12 W24 W48
  The SAS is a self-report inventory of anxiety symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Jindong Chen, MD, Study Director — Second Xiangya Hospital of Central South University
Locations (1):
- Mental Health Institute, Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
June 1,2020, Email to Dr. Chen Jindong(chenjd269@163.com)

REFERENCES:
- [Background] Kessler RC, Birnbaum H, Bromet E, Hwang I, Sampson N, Shahly V. Age differences in major depression: results from the National Comorbidity Survey Replication (NCS-R). Psychol Med. 2010 Feb;40(2):225-37. doi: 10.1017/S0033291709990213. Epub 2009 Jun 17. PMID 19531277
- [Background] Monroe SM, Harkness KL. Recurrence in major depression: a conceptual analysis. Psychol Rev. 2011 Oct;118(4):655-74. doi: 10.1037/a0025190. PMID 21895384
- [Background] Appleton KM, Rogers PJ, Ness AR. Updated systematic review and meta-analysis of the effects of n-3 long-chain polyunsaturated fatty acids on depressed mood. Am J Clin Nutr. 2010 Mar;91(3):757-70. doi: 10.3945/ajcn.2009.28313. Epub 2010 Feb 3. PMID 20130098
- [Background] McNamara RK, Carlson SE. Role of omega-3 fatty acids in brain development and function: potential implications for the pathogenesis and prevention of psychopathology. Prostaglandins Leukot Essent Fatty Acids. 2006 Oct-Nov;75(4-5):329-49. doi: 10.1016/j.plefa.2006.07.010. Epub 2006 Sep 1. PMID 16949263
- [Background] Freeman MP, Rapaport MH. Omega-3 fatty acids and depression: from cellular mechanisms to clinical care. J Clin Psychiatry. 2011 Feb;72(2):258-9. doi: 10.4088/JCP.11ac06830. No abstract available. PMID 21382308
- [Background] Bloch MH, Hannestad J. Omega-3 fatty acids for the treatment of depression: systematic review and meta-analysis. Mol Psychiatry. 2012 Dec;17(12):1272-82. doi: 10.1038/mp.2011.100. Epub 2011 Sep 20. PMID 21931319
- [Background] Sprecher H. Metabolism of highly unsaturated n-3 and n-6 fatty acids. Biochim Biophys Acta. 2000 Jul 19;1486(2-3):219-31. doi: 10.1016/s1388-1981(00)00077-9. No abstract available. PMID 10903473
- [Background] Xie L, Innis SM. Association of fatty acid desaturase gene polymorphisms with blood lipid essential fatty acids and perinatal depression among Canadian women: a pilot study. J Nutrigenet Nutrigenomics. 2009;2(4-5):243-50. doi: 10.1159/000255636. Epub 2010 Apr 15. PMID 20395685
- [Background] Lalovic A, Klempan T, Sequeira A, Luheshi G, Turecki G. Altered expression of lipid metabolism and immune response genes in the frontal cortex of suicide completers. J Affect Disord. 2010 Jan;120(1-3):24-31. doi: 10.1016/j.jad.2009.04.007. PMID 19443042
- [Derived] Wang F, Yuan H, Jin K, Tang H, Guo J, Wang CY, Chen J, Dong F, Wang L. Effects of fish oil supplementation on bone turnover markers in depression: a pilot study. Front Nutr. 2024 Dec 12;11:1464526. doi: 10.3389/fnut.2024.1464526. eCollection 2024. PMID 39726877
- [Derived] Yang R, Wang L, Jin K, Cao S, Wu C, Guo J, Chen J, Tang H, Tang M. Omega-3 Polyunsaturated Fatty Acids Supplementation Alleviate Anxiety Rather Than Depressive Symptoms Among First-Diagnosed, Drug-Naive Major Depressive Disorder Patients: A Randomized Clinical Trial. Front Nutr. 2022 Jul 12;9:876152. doi: 10.3389/fnut.2022.876152. eCollection 2022. PMID 35903448
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03295708/Prot_SAP_000.pdf